CLINICAL TRIAL: NCT02793635
Title: Impact of Gait Training With an Exoskeleton on Walking Function After Spinal Cord Injury (SCI)
Brief Title: Indego Exoskeleton After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Hannifin Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-01399
Record Dates: First submitted 2016-05-24; First posted 2016-06-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injury
Keywords: Paraplegia; Gait; Exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCI Patients (Experimental): * 10 subjects with complete or incomplete SCI (> 1 year post-injury) with preserved LE function will be recruited.
  * No control group
  Interventions: Device: Indego Powered Exoskeleton

INTERVENTIONS:
Device: Indego Powered Exoskeleton — Subjects who have Spinal Cord Injury will wear the Indego device which will include being trained and evaluated for fifteen (15) sessions.
  Other Names: Vanderbilt exoskeleton

SUMMARY:
The purpose of this study is to assess the use of Indego as a gait training tool for subjects with complete or incomplete paraplegia as a result of spinal cord injury (SCI) who have preserved lower extremity function. It is hypothesized that subjects with complete or incomplete paraplegia who have preserved their lower extremity function will experience functional improvements after gait training with the Indego exoskeleton.

Subjects will complete a total of fifteen (15) sessions which include a combination of the following; Physical Therapy Evaluation, Indego Training, Mid-Way Assessment, and Post-Assessment.

The aim of this study is to measure the impact of gait training with the Indego device on body structure, function, and participation. Additionally it will assess the perceptions of physical therapists and subjects with SCI on the effectiveness of gait training with the Indego exoskeleton in subjects with preserved limited function.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Height 5'1" to 6'3" (Acceptable height may vary by a few inches depending on femur length)
* Weight 250 lbs or less
* Present with paraplegia resulting from a complete or incomplete (AIS A, B, C, or D) Spinal Cord Injury (>1 year post-injury), with preserved LE function
* Uses wheelchair as primary means of mobility in the community
* Able to ambulate 14 meters with assist of 2 people and no orthostasis. Subjects may use any combination of stability aids and/or bracing.
* Medical clearance for weight bearing and locomotor training

  * Bone density exams will be at the discretion of each sites' Principle Investigator
* Passive range of motion (PROM) at shoulders, trunk, hips, knees and ankles within functional limits for safe gait and use of appropriate assistive device/stability aid
* Skin intact where interfaces with the Indego device
* Modified Ashworth Scale 3 or less in bilateral LEs
* Blood pressure and heart rate within Locomotor Training Guidelines

  * At rest: Systolic 150 or less Diastolic 90 or less and Heart rate 105 or less
  * Exercise: Systolic 180 or less Diastolic 105 or less and Heart Rate 145 or less

Exclusion Criteria:

* Inability to meet ALL inclusion criteria
* Currently participating in physical therapy for gait training
* Joint contractures of the shoulders, trunk, hips knees or ankles deemed unsafe for locomotor training by PT and or MD
* Edema that would put skin at risk for breakdown
* Modified Ashworth Spasticity of 4
* Inability to achieve adequate fit of the Indego device
* Pregnancy
* Colostomy bag

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Functional ambulation category (FAC) to measure gait quality | 1 Day
  Categorizes patients according to basic motor skills necessary for functional ambulation
10 Meter Walking Test to measure fast gait speed | 1 Day
  Assesses walking speed in meters per second over a short duration
6 Minute Walking test to measure endurance | 6 Minutes
  Measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Charles Hospital, Port Jefferson, New York
  - TIRR Memorial Hermann, Houston, Texas
  - Sheltering Arms, Mechanicsville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided